CLINICAL TRIAL: NCT01729156
Title: Effects of Metformin on Hepatic Free Fatty Acid Metabolism in Patients Diagnosed With Type 2 Diabetes: A C11 PET Study
Brief Title: Effects of Metformin on Hepatic FFA Metabolism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lars Christian Gormsen (Other)
Responsible Party: Sponsor-Investigator, Lars Christian Gormsen, Senior Registrar, MD PhD, Aarhus University Hospital
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: C11palmitatMetformin
Record Dates: First submitted 2012-11-13; First posted 2012-11-20 (Estimated); Results first posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-09

CONDITIONS: Type 2 Diabetes; Dyslipidemia
Keywords: Type 2 diabetes; Hepatic fatty acid oxidation; Dyslipidemia; Metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Dyslipidemias | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Healthy controls (Other): Healthy controls receiving 1000 mg metformin twice daily for 3 months
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Metformin (Active Comparator): Metformin "Sandoz", 1000 mg twice daily for 3 months
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — 1000 mg metformin twice daily in 3 months
  Other Names: Metformin "Sandoz" 500 mg
  Arms: Healthy controls; Metformin
Drug: Placebo — 2 tablets twice daily in 3 months
  Arms: Placebo

SUMMARY:
Background: Metformin treatment has beneficial effects on both glucose and lipid metabolism. Whereas there is general agreement that the blood glucose lowering effect of metformin results from inhibition of hepatic gluconeogenesis, it is less clear exactly how the drug lowers blood triglyceride concentration. There are indications that it enhances hepatic free fatty acid (FFA) oxidation thus diminishing substrate for reesterification and resecretion as very-low-density-lipoprotein (VLDL) triglycerides (TG). However, the liver is not easily accessible for sampling in humans and data on the clinical effects of metformin in the liver are therefore lacking. This may change due to the increasing use of the positron emission tomography (PET) technique. Using PET isotopes (11C or 18F) coupled to either palmitate or a fatty acid analogue, it is possible to non-invasively measure hepatic fatty acid handling.

Aim: To determine how 3 months metformin treatment (1000 mg twice daily) affects hepatic lipid and glucose metabolism in patients with newly diagnosed type 2 diabetes.

Design: Randomized, placebo controlled, double-blind parallel study with patients receiving either metformin or placebo. A control group of BMI and age-matched non-diabetic individuals will receive metformin for 3 months.

Hypothesis: Metformin lowers VLDL-TG secretion and circulating triglycerides by increasing hepatic fatty acid oxidation

ELIGIBILITY:
Inclusion Criteria:

* Recently diagnosed type 2 diabetes
* Age 50-70 years
* BMI<40

Exclusion Criteria:

* Insulin treatment
* NASH (non alcoholic steatohepatitis)
* Cancer
* Anemia
* HbA1C>8.5 %
* Chronic or acute pancreatitis
* Alcohol or medicine abuse
* Allergy towards metformin
* Claustrophobia
* Severe obesity (weight >130 kilogram)

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-01; Primary Completion 2017-05-05 (Actual); Study Completion 2017-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars C Gormsen, MD PhD, Principal Investigator — Aarhus University Hospital

REFERENCES:
- [Derived] Gormsen LC, Sondergaard E, Christensen NL, Brosen K, Jessen N, Nielsen S. Metformin increases endogenous glucose production in non-diabetic individuals and individuals with recent-onset type 2 diabetes. Diabetologia. 2019 Jul;62(7):1251-1256. doi: 10.1007/s00125-019-4872-7. Epub 2019 Apr 11. PMID 30976851

RESULTS

PARTICIPANT FLOW:
Groups:
- Metformin: Metformin "Teva", 1000 mg twice daily for 3 months
  Metformin: 1000 mg metformin twice daily in 3 months
Period: Overall Study
Arm/Group | Healthy Controls | Placebo | Metformin
Started | 12 | 12 | 12
Completed | 11 | 12 | 12
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Controls | Placebo | Metformin | Total
Number analyzed (Participants) | 12 | 12 | 12 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (6) | 60 (5) | 64 (5) | 62 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 6 | 15
  Male | 6 | 9 | 6 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 12 | 12 | 12 | 36
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m2] | 27.3 (4.1) | 31.2 (4.3) | 30.3 (5.7) | 29.6 (4.7)
HbA1C [Mean (Standard Deviation); unit: mmol/mmol] | 37 (3) | 45 (6) | 51 (6) | 44 (5)

OUTCOME MEASURES:

1. Primary Outcome: Hepatic Fatty Acid Oxidation
Description: Hepatic fatty acid oxidation assessed by dynamic C11-palmitate PET
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: micromol/ml/min
Arm/Group | Healthy Controls | Placebo | Metformin
Number analyzed (Participants) | 10 | 11 | 10
micromol/ml/min | 0.052 (0.024) | 0.045 (0.024) | 0.042 (0.017)

2. Primary Outcome: Hepatic Fatty Acid Reesterification
Description: Hepatic fatty acid reesterification assessed by C11-palmitate PET
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: micromol/ml/min
Arm/Group | Healthy Controls | Placebo | Metformin
Number analyzed (Participants) | 10 | 11 | 10
micromol/ml/min | 0.134 (0.056) | 0.091 (0.035) | 0.113 (0.025)

3. Primary Outcome: Hepatic Fatty Acid Uptake
Description: Hepatic fatty acid uptake assessed by C11-palmitate PET
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: micromol/ml/min
Arm/Group | Healthy Controls | Placebo | Metformin
Number analyzed (Participants) | 10 | 11 | 10
micromol/ml/min | 0.186 (0.067) | 0.137 (0.051) | 0.155 (0.029)

4. Primary Outcome: VLDL-TG Secretion
Description: Hepatic VLDL-TG secretion assessed by [1-14C] VLDL tracer
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: micromol/min
Arm/Group | Healthy Controls | Placebo | Metformin
Number analyzed (Participants) | 11 | 11 | 11
micromol/min | 48 (30) | 83 (49) | 71 (31)

5. Primary Outcome: Whole Body Glucose Rd
Description: Whole body basal glucose metabolism assessed by [3-3H]glucose tracer kinetics
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mg/kg/min
Arm/Group | Healthy Controls | Placebo | Metformin
Number analyzed (Participants) | 11 | 12 | 11
mg/kg/min | 1.74 (0.29) | 1.30 (0.31) | 1.78 (0.43)

6. Secondary Outcome: Fatty Acid Turnover
Description: Fatty acid turnover assessed as whole body C11-palmitate turnover
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: micromol/min
Arm/Group | Healthy Controls | Placebo | Metformin
Number analyzed (Participants) | 10 | 11 | 11
micromol/min | 464 (127) | 476 (149) | 559 (295)

7. Secondary Outcome: VLDL-TG Oxidation
Description: VLDL-TG oxidation assessed by 14C carbon dioxide (CO2) in exhaled breath
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: percentage of 14C-VLDL
Arm/Group | Healthy Controls | Placebo | Metformin
Number analyzed (Participants) | 11 | 12 | 11
percentage of 14C-VLDL | 29 (5) | 30 (7) | 27 (9)

ADVERSE EVENTS:
Time Frame: During the 90 days trial
Arm/Group | Healthy Controls | Placebo | Metformin
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 1/12 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Controls (N=12) | Placebo (N=12) | Metformin (N=12)
Gastrointestinal uncomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fractured vertebral column (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2013-02-04): https://cdn.clinicaltrials.gov/large-docs/56/NCT01729156/Prot_000.pdf